CLINICAL TRIAL: NCT04144803
Title: Brain Oxygenation During Prehospital Anesthesia: an Observational Study (The BOPRA Study)
Brief Title: Brain Oxygenation During Prehospital Anesthesia: an Observational Study
Acronym: BOPRA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: FinnHEMS Ltd (Unknown); Turku University Hospital (Other Government); Tampere University Hospital (Other); Oulu University Hospital (Other); Lapland Hospital District (Unknown); Kuopio University Hospital (Other); Metropolia University of Applied Sciences (Other); Turku University of Applied Sciences (Unknown); Tampere University (Other); Oulu University of Applied Sciences (Unknown); Savonia University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Jouni Nurmi, MD, associate professor, Helsinki University Central Hospital
Other Study IDs: BOPRA
Record Dates: First submitted 2019-10-07; First posted 2019-10-30 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Critically Ill; Major Trauma; Anesthesia; Emergencies
MeSH Terms: conditions — Critical Illness; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral desaturation group: absolute drop of forehead cerebral oxygen saturation ≥ 10% from baseline for ≥ 5 minutes during prehospital anesthesia
  Interventions: Diagnostic Test: Cerebral near-infrared spectroscopy
- Control group: no absolute drop of forehead cerebral oxygen saturation ≥ 10% from baseline for ≥ 5 minutes during prehospital anesthesia
  Interventions: Diagnostic Test: Cerebral near-infrared spectroscopy

INTERVENTIONS:
Diagnostic Test: Cerebral near-infrared spectroscopy — Nonin H500 one-channel near-infrared spectroscopy monitor on forehead of the patient from before induction of anesthesia to arrival to hospital

SUMMARY:
Brain oxygenation of adult patients undergoing prehospital emergency anesthesia is monitored using noninvasive near-infrared spectroscopy. Patients are afterwards interviewed to define neurological outcome to measure quality of life. The purpose of this study is to reveal the risk factors of prehospital anesthesia related cerebral desaturation events (CDE) and to define the association between CDE and survival, neurological outcome or quality of life.

ELIGIBILITY:
Inclusion Criteria:

* sedation or anesthesia provided to facilitate endotracheal intubation, performed by Helicopter Emergency Medical Services (HEMS) team regardless of the reason

Exclusion Criteria:

* Ongoing cardiopulmonary resuscitation at the time of intubation
* Physical barrier for near-infrared spectroscopy measuring (e.g. forehead laceration)
* HEMS unit does not escort patient to the hospital (exception: in case of death on scene after inclusion, patient is included)
* Workload too high to ensure standard level of clinical care during the study
* For interviews: no competence in Finnish, Swedish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing prehospital anesthesia and endotracheal intubation regardless of indication
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Favorable neurological outcome | 30 days
  modified Rankin scale ≤2 (scale 0-6, 0 asymptomatic, 6 expired)
Cerebral desaturation event | through prehospital care, approximately 60 minutes
  an absolute drop of forehead cerebral saturation ≥ 10% from baseline for ≥ 5 minutes

SECONDARY OUTCOMES:
Survival | 30 days
  Survival
Survival | 365 days
  Survival
Favorable neurological outcome | 1 year
  modified Rankin scale ≤2 (scale 0-6, 0 asymptomatic, 6 expired)
15D score | 1 year
  Heal-Related Quality of Life measured using 15-D instrument, scale 0-1 (0 = being dead, 0.0162 = being unconscious or comatose, 1 = no problems on any dimension = 'full' HRQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Jouni Nurmi, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (6):
- Finland (6):
  - FinnHEMS 60 / Kuopio University Hospital, Kuopio
  - FinnHEMS 50 / Oulu University Hospital, Oulu
  - FinnHEMS 51 / Lapland hospital district, Rovaniemi
  - FinnHEMS 30 / Tampere University Hospital, Tampere
  - FinnHEMS 20 / Turku University Hospital, Turku
  - FinnHEMS 10 / Helsinki University Hospital, Vantaa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saviluoto A, Raatiniemi L, Makela S, Toivonen T, Setala P, Kirves H, Tommila M, Toivonen P, Tukia S, Nurmi J. Association of Cerebral Oxygenation During Prehospital Anaesthesia and Functional Outcome: A Prospective, Observational Multi-Centre Cohort Study of 1014 Patients. Acta Anaesthesiol Scand. 2026 Jan;70(1):e70161. doi: 10.1111/aas.70161. PMID 41359999